CLINICAL TRIAL: NCT01669486
Title: The Pain in Intensive Care Unit: An Experimental Research to Compare Behavioural Pain Scale (BPS) and Critical Care Pain Observation Tool (CPOT)
Brief Title: The Pain in Intensive Care Unit: Different Rating System Comparing
Acronym: ICPain
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Paolo Severgnini, Prof., Università degli Studi dell'Insubria
Other Study IDs: 1514
Record Dates: First submitted 2012-06-14; First posted 2012-08-21 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Critical Illness
Keywords: Pain; ICU; Mechanical ventilation; CPOT; BPS
MeSH Terms: conditions — Critical Illness; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICU patients: All patients admitted to ICU for a minimal hospitalization of 24 hours, invasive mechanically ventilated, will be evaluated with CPOT and BPS scores, during nurses work, in particular before and after nurses manoeuvers.
  Interventions: Other: CPOT, BPS

INTERVENTIONS:
Other: CPOT, BPS — Scoring pain of the patients during nurses activity in ICU, in particular before and after nurses manoeuvers.

SUMMARY:
The purpose of this research is to find the best system for assessing the pain of critically ill patient in Intensive Care Unit (ICU).

At first the investigators assess the sedation of the patient with the scale sedation-agitation scale (SAS) or the delirium with the confusion assessment method, if the patient is too sedated or delirious the investigators consider him unable to use the Visual Analogic Scale (VAS).

The investigators compare two different scales Critical Care Pain Observation Tool (CPOT) and Behavioural Pain Scale (BPS) which include no verbal items. Each items has been evaluated in three different moments: before, during and after the nurses' care.

The investigators compare the scales between them. Then, every time the investigators value the score of these scales with the self-report of patients with the VAS scale (when it is possible) and finally with the physiological parameters (blood pressure, heart rate and respiratory rate).

In the end, the investigators compare two different classes of patient: the surgical and medical one. The investigators search for some differences in the perception of the pain between these two classes.

DETAILED DESCRIPTION:
This study has specific aims:

1. to find the best method to evaluate the pain in critically ill patients;
2. to compare the perception of pain analysed trough CPOT and BPS;
3. to compare CPOT and BPS between medical and surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* require of Mechanical Ventilation (MV)
* Hospitalization on ICU > 24 hours

Exclusion Criteria:

* Age < 18 years
* Tetraplegic
* Neuromuscolar disease
* Neuromuscolar blocking agents by continuous infusion
* Spontaneous breathing without Mechanical Ventilation (MV)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female Critically ill patients Mechanically ventilated patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The evaluation of pain in critically ill patients | Participants will be followed for 3 days
  The measurement of pain with no verbal items of different pain scales: facial expression, movements of the body, muscle tone, compliance of mechanical ventilation, movements of the arms. We'll evaluate the level of pain before and after nurses manoeuvers

SECONDARY OUTCOMES:
The comparisation beetween the CPOT and the BPS scales | Participants will be followed for 3 days
  The comparisation beetween the different items of two scales: CPOT (facial expression, movements of the body, muscle tone, compliance of mechanical ventilation) and BPS (facial expression, movements of the arms, compliance of mechanical ventilation).
The comparisation of CPOT and BPS between medical and surgical critically ill patients | Participants will be followed for 3 days
  We'll measure facial expression, movements of the body, muscle tone, compliance of mechanical ventilation, movements of the arms, according with BPS and CPOT scores in two classes of patient: the surgical and medical critically ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo MD Severgnini, Prof., Study Director — Universita' degli Studi dell'Insubria, Varese, Italy
Locations (1):
- Azienda ospedaliera ospedale Circolo e Fondazione Macchi, Varese, Varese, Italy

REFERENCES:
- [Derived] Severgnini P, Pelosi P, Contino E, Serafinelli E, Novario R, Chiaranda M. Accuracy of Critical Care Pain Observation Tool and Behavioral Pain Scale to assess pain in critically ill conscious and unconscious patients: prospective, observational study. J Intensive Care. 2016 Nov 7;4:68. doi: 10.1186/s40560-016-0192-x. eCollection 2016. PMID 27833752